CLINICAL TRIAL: NCT03599622
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of BMS-986165 in Subjects With Moderate to Severe Crohn's Disease
Brief Title: An Investigational Study of Experimental Medication BMS-986165 in Participants With Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated because of lack of efficacy in the short term acute phase
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-023; 2017-001976-48 (EudraCT Number)
Record Dates: First submitted 2018-07-11; First posted 2018-07-26 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Granulomatous Colitis; Crohn's Disease; Crohn's Enteritis; Granulomatous Enteritis
MeSH Terms: conditions — Crohn Disease | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986165 Dose 1 (Experimental)
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 2 (Experimental)
  Interventions: Drug: BMS-986165
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: BMS-986165 Dose 1; BMS-986165 Dose 2
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of BMS-986165 compared to placebo in participants with moderately to severely active Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Crohn's Disease (CD) for at least 3 months prior to screening, including ileal, colonic, or ileo-colonic disease distribution
* Must have had an inadequate response, loss of response, or intolerance to 1 or more of the standard treatments
* Must have active moderate to severe CD
* Men and women must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Severe or fulminant colitis that is likely to require surgery or hospitalization
* Presence of a diagnosis of alternative forms of colitis (infectious, inflammatory including ulcerative colitis, malignant, toxic, indeterminate, etc.) other than Crohn's Disease
* Previous exposure to BMS-986165 in any study
* Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, immunologic, psychiatric, or local active infection/infectious illness) that, in the investigator's judgment, will substantially increase the risk to the participant

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (259):
- United States (52):
  - Local Institution - 0258, Los Angeles, California
  - Local Institution - 0247, Aurora, Colorado
  - Local Institution - 0001, Hamden, Connecticut
  - Local Institution - 0255, Clearwater, Florida
  - Local Institution - 0259, Jacksonville, Florida
  - Local Institution - 0261, Jacksonville, Florida
  - Local Institution - 0276, Largo, Florida
  - Local Institution - 0232, Miami, Florida
  - Local Institution - 0162, New Port Richey, Florida
  - Local Institution - 0201, Orlando, Florida
  - Local Institution - 0249, Orlando, Florida
  - Local Institution - 0166, Tampa, Florida
  - Local Institution - 0248, Zephyrhills, Florida
  - Local Institution - 0277, Suwanee, Georgia
  - Local Institution - 0358, Suwanee, Georgia
  - Local Institution - 0319, Chicago, Illinois
  - Local Institution - 0346, Glenview, Illinois
  - Local Institution - 0301, Indianapolis, Indiana
  - Local Institution - 0253, Iowa City, Iowa
  - Local Institution - 0282, Shreveport, Louisiana
  - Local Institution - 0003, Chesterfield, Michigan
  - Local Institution - 0218, Chesterfield, Michigan
  - Local Institution - 0047, Wyoming, Michigan
  - Local Institution - 0223, Ypsilanti, Michigan
  - Local Institution - 0231, Jackson, Mississippi
  - Local Institution - 0156, Ocean Springs, Mississippi
  - Local Institution - 0359, St Louis, Missouri
  - Local Institution - 0011, Las Vegas, Nevada
  - Local Institution - 0043, Lake Success, New York
  - Local Institution - 0308, New York, New York
  - Local Institution - 0226, Monroe, North Carolina
  - Local Institution - 0349, Oklahoma City, Oklahoma
  - Local Institution - 0238, Hershey, Pennsylvania
  - Local Institution - 0125, Pittsburgh, Pennsylvania
  - Local Institution - 0122, Sayre, Pennsylvania
  - Local Institution - 0357, Wyomissing, Pennsylvania
  - Local Institution - 0105, Charleston, South Carolina
  - Local Institution - 0072, Nashville, Tennessee
  - Local Institution - 0264, Arlington, Texas
  - Local Institution - 0246, Garland, Texas
  - Local Institution - 0252, San Antonio, Texas
  - Local Institution - 0307, San Antonio, Texas
  - Local Institution - 0073, Southlake, Texas
  - Local Institution - 0240, Spring, Texas
  - Local Institution - 0302, Tyler, Texas
  - Local Institution, Lynchburg, Virginia
  - Local Institution - 0224, Richmond, Virginia
  - Local Institution - 0327, Seattle, Washington
  - Local Institution - 0266, Seattle, Washington
  - Local Institution - 0191, Seattle, Washington
  - Local Institution - 0331, Vancouver, Washington
  - Local Institution - 0356, Milwaukee, Wisconsin
- Australia (9):
  - Local Institution - 0268, South Brisbane, Queensland
  - Local Institution - 0254, Woolloongabba, Queensland
  - Local Institution - 0265, Adelaide, South Australia
  - Local Institution - 0289, Woodville, South Australia
  - Local Institution - 0042, Ballarat, Victoria
  - Local Institution - 0041, Clayton, Victoria
  - Local Institution - 0040, Melbourne, Victoria
  - Local Institution - 0351, Melbourne, Victoria
  - Local Institution - 0275, Murdoch, Western Australia
- Belgium (4):
  - Local Institution - 0316, Antwerp
  - Local Institution - 0305, Edegem
  - Local Institution - 0322, Ghent
  - Local Institution - 0314, Yvoir
- Brazil (9):
  - Local Institution - 0256, Salvador, Estado de Bahia
  - Local Institution - 0262, Salvador, Estado de Bahia
  - Local Institution - 0069, Juiz de Fora, Minas Gerais
  - Local Institution - 0086, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0058, Botucato, São Paulo
  - Local Institution - 0059, Santo André, São Paulo
  - Local Institution - 0045, São Bernardo do Campo, São Paulo
  - Local Institution - 0085, São José do Rio Preto, São Paulo
  - Local Institution - 0017, Rio de Janeiro
- Canada (8):
  - Local Institution - 0048, Calgary, Alberta
  - Local Institution - 0324, Edmonton, Alberta
  - Local Institution - 0300, Edmonton, Alberta
  - Local Institution - 0159, Vancouver, British Columbia
  - Local Institution - 0283, Etobicoke, Ontario
  - Local Institution - 0312, London, Ontario
  - Local Institution - 0236, Toronto, Ontario
  - Local Institution - 0317, Montreal, Quebec
- China (10):
  - Local Institution - 0280, Xiamen, Fujian
  - Local Institution - 0225, Guangzhou, Guangdong
  - Local Institution - 0228, Guangzhou, Guangdong
  - Local Institution - 0221, Changsha, Hunan
  - Local Institution - 0220, Nanjing, Jiangsu
  - Local Institution - 0306, Nanjing, Jiangsu
  - Local Institution - 0250, Changchun, Jilin
  - Local Institution - 0299, Shenyang, Liaoning
  - Local Institution - 0219, Shanghai, Shanghai Municipality
  - Local Institution - 0234, Shanghai, Shanghai Municipality
- Czechia (7):
  - Local Institution - 0337, Brno
  - Local Institution - 0360, Brno
  - Local Institution - 0057, Hradec Králové
  - Local Institution - 0352, Ostrava
  - Local Institution - 0071, Ostrava
  - Local Institution - 0350, Pardubice
  - Local Institution - 0075, Prague
- Denmark (3):
  - Local Institution - 0192, Aalborg
  - Local Institution - 0202, Copenhagen NV
  - Local Institution - 0320, Odense
- France (6):
  - Local Institution - 0110, Clichy
  - Local Institution - 0168, Colombes
  - Local Institution - 0343, Montpellier
  - Local Institution - 0084, Saint-Etienne
  - Local Institution - 0127, Toulouse
  - Local Institution - 0167, Toulouse
- Germany (14):
  - Local Institution - 0099, Berlin
  - Local Institution - 0090, Berlin
  - Local Institution - 0339, Brandenburg
  - Local Institution - 0212, Frankfurt
  - Local Institution - 0178, Halle
  - Local Institution, Halle
  - Local Institution - 0294, Hanover
  - Local Institution - 0089, Jena
  - Local Institution - 0190, Kiel
  - Local Institution - 0321, Mannheim
  - Local Institution - 0140, Münster
  - Local Institution - 0257, Regensburg
  - Local Institution - 0340, Tübingen
  - Local Institution - 0102, Ulm
- Hungary (11):
  - Local Institution - 0104, Békéscsaba
  - Local Institution - 0242, Budapest
  - Local Institution - 0263, Budapest
  - Local Institution - 0211, Budapest
  - Local Institution - 0100, Budapest
  - Local Institution - 0292, Budapest
  - Local Institution - 0054, Debrecen
  - Local Institution - 0083, Gyöngyös
  - Local Institution - 0210, Mohács
  - Local Institution - 0243, Szeged
  - Local Institution - 0164, Vác
- Ireland (5):
  - Local Institution - 0348, Tallaght, Dublin
  - Local Institution - 0335, Ballinasloe, Galway
  - Local Institution - 0336, Drogheda, Louth
  - Local Institution - 0330, Dublin
  - Local Institution - 0332, Galway
- Israel (4):
  - Local Institution - 0197, Beersheba
  - Local Institution - 0186, Nahariya
  - Local Institution - 0184, Petah Tikva
  - Local Institution - 0198, Rehovot
- Italy (14):
  - Local Institution - 0290, Bologna
  - Local Institution - 0298, Castellana Grotte
  - Local Institution - 0171, Catanzaro
  - Local Institution - 0056, Messina
  - Local Institution - 0304, Milan
  - Local Institution - 0115, Milan
  - Local Institution - 0311, Milan
  - Local Institution - 0297, Monserrato
  - Local Institution - 0310, Negrar
  - Local Institution - 0128, Padua
  - Local Institution - 0170, Pavia
  - Local Institution - 0161, Roma
  - Local Institution - 0119, Rozzano
  - Local Institution - 0285, Torino
- Japan (24):
  - Local Institution - 0182, Toyoake, Aichi-ken
  - Local Institution - 0199, Hirosaki, Aomori
  - Local Institution - 0205, Sakura-shi, Chiba
  - Local Institution - 0328, Tōon, Ehime
  - Local Institution - 0326, Fukui-shi, Fukui
  - Local Institution - 0204, Chikushino-shi, Fukuoka
  - Local Institution - 0187, Kurume-shi, Fukuoka
  - Local Institution - 0323, Sapporo, Hokkaido
  - Local Institution - 0217, Sapporo, Hokkaido
  - Local Institution - 0183, Nishinomiya, Hyōgo
  - Local Institution - 0207, Sagamihara-shi, Kanagawa
  - Local Institution - 0200, Sendai, Miyagi
  - Local Institution - 0194, Omura-shi, Nagasaki
  - Local Institution - 0318, Urasoe-Shi, Okinawa
  - Local Institution - 0179, Suita-shi, Osaka
  - Local Institution - 0185, Ōtsu, Shiga
  - Local Institution - 0189, Hamamatsu, Shizuoka
  - Local Institution - 0213, Bunkyo-ku, Tokyo
  - Local Institution - 0195, Minato-ku, Tokyo
  - Local Institution - 0188, Hiroshima
  - Local Institution - 0206, Kyoto
  - Local Institution - 0214, Miyazaki
  - Local Institution - 0196, Saga
  - Local Institution - 0203, Sapporo
- Mexico (5):
  - Local Institution - 0106, Guadalajara, Jalisco
  - Local Institution - 0007, Mexico City, Mexico City
  - Local Institution - 0009, Cuernavaca, Morelos
  - Local Institution - 0109, Monterrey, Nuevo León
  - Local Institution - 0029, Querétaro
- Local Institution - 0303, Amsterdam, Netherlands
- Poland (16):
  - Local Institution - 0245, Bydgoszcz
  - Local Institution - 0177, Bydgoszcz
  - Local Institution - 0065, Krakow
  - Local Institution - 0284, Lodz
  - Local Institution - 0098, Lodz
  - Local Institution - 0291, Lublin
  - Local Institution - 0278, Nowy Targ
  - Local Institution - 0176, Olsztyn
  - Local Institution - 0082, Sopot
  - Local Institution - 0063, Tychy
  - Local Institution - 0271, Warsaw
  - Local Institution - 0288, Warsaw
  - Local Institution - 0026, Warsaw
  - Local Institution - 0279, Warsaw
  - Local Institution - 0160, Wroclaw
  - Local Institution - 0034, Wroclaw
- Portugal (2):
  - Local Institution - 0174, Guimarães
  - Local Institution - 0216, Santa Maria da Feira
- Romania (6):
  - Local Institution - 0067, Bucharest
  - Local Institution - 0044, Bucharest
  - Local Institution - 0163, Bucharest
  - Local Institution - 0074, Bucharest
  - Local Institution - 0005, Timișoara
  - Local Institution - 0060, Timișoara
- Russia (14):
  - Bioterm, Barnaul
  - Hospital Irkutsk Scientific Center, Irkutsk
  - Republican Clinical Hospital Ministry of Health Republic of Tatarstan, Kazan'
  - City Clinical Hospital Number 24, Moscow
  - Medical Center SibNovoMed, Novosibirsk
  - Novosibirsk Gastrocenter, Novosibirsk
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Medical Center Healthy Family, Novosibirsk
  - Clinic Ultrasound 4D, Pyatigorsk
  - Saint Petersburg State Budgetary Institution of Health City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - Tomsk Regional Clinical Hospital, Tomsk
  - Multidisciplinary Consultative and Diagnostic Center, Tyumen
  - Novgorod Regional Clinical Hospital, Veliky Novgorod
- South Korea (10):
  - Local Institution - 0046, Seongnam-si, Gyeonggi-do
  - Local Institution - 0158, Ansan-si
  - Local Institution - 0149, Busan
  - Local Institution - 0064, Daegu
  - Local Institution - 0061, Daegu
  - Local Institution - 0150, Incheon
  - Local Institution - 0015, Seoul
  - Local Institution - 0016, Seoul
  - Local Institution - 0012, Wŏnju
  - Local Institution - 0032, Yangsan
- Spain (12):
  - Local Institution - 0329, Alicante
  - Local Institution - 0274, Barcelona
  - Local Institution - 0154, Fuenlabrada
  - Local Institution - 0080, Girona
  - Local Institution - 0021, Las Palmas de Gran Canaria
  - Local Institution, LHospitalet de Llobregat
  - Local Institution - 0325, Sabadell
  - Local Institution - 0113, Santander
  - Local Institution - 0309, Santiago de Compostelle
  - Local Institution - 0313, Seville
  - Local Institution - 0107, Seville
  - Local Institution - 0004, Valencia
- Local Institution - 0180, Bern, Switzerland
- Taiwan (4):
  - Local Institution - 0173, Kaohsiung City
  - Local Institution - 0148, Taichung
  - Local Institution - 0267, Taipei
  - Local Institution - 0152, Taoyuan District
- United Kingdom (8):
  - Local Institution - 0341, Birmingham
  - Local Institution - 0144, Blackpool
  - Local Institution - 0235, Cambridge
  - Local Institution - 0354, Cannock
  - Local Institution - 0165, Cheshire
  - Local Institution - 0157, Glasgow
  - Local Institution - 0353, Manchester
  - Local Institution - 0208, Swansea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study has a treat-through design
Pre-assignment Details: Enrollment into the 12 mg BMS-986165 arm was discontinued. Participants who were randomized to 12 mg BMS-986165 continued on their originally assigned double-blind study treatment. These participants completed all study procedures and assessments outlined in the current version of the protocol.
Groups:
- Placebo: Placebo was taken twice per day over 12 weeks. Participants who achieved a clinical response after week 12 continued to take placebo twice daily until the end of week 52. Participants who did not achieve clinical response at week 12 but had an appropriate safety profile were eligible to receive open-label BMS-986165 6 mg twice per day until week 52. Week 12 responders (Placebo) and week 12 non-responders (BMS-986165 6 mg OL) who continued to derive a clinical benefit from their respective treatments at week 26/52 and week 52 respectively were eligible to receive BMS-986165 6 mg twice daily for up week 104.
- 3 mg BMS-986165: BMS-986165 3 mg was taken orally twice per day over 12 weeks. Participants who achieved a clinical response after the week 12 continued to take BMS-986165 3 mg orally twice daily until the end of week 52. Participants who did not achieve clinical response at week 12 but had an appropriate safety profile were eligible to receive BMS-986165 6 mg twice per day until week 52. Week 12 responders (BMS-986165 3 mg) and week 12 non-responders (BMS-986165 6 mg OL) who continued to derive a clinical benefit from their respective treatments at week 26/52 and week 52 respectively were eligible to receive open label BMS-986165 6 mg twice daily for up to week 104.
- 6 mg BMS-986165: BMS-986165 6 mg was taken orally twice per day over 12 weeks. Participants who achieved a clinical response after the week 12 continued to take BMS-986165 6 mg orally twice daily until the end of week 52. Participants who did not achieve clinical response at week 12 but had an appropriate safety profile were eligible to receive BMS-986165 6 mg twice per day until week 52. Week 12 responders and week 12 non-responders who continued to derive a clinical benefit from their respective treatments at week 26/52 and week 52 respectively were eligible to receive open label BMS-986165 6 mg twice daily up to week 104.
- 12 mg BMS-986165: BMS-986165 12 mg was taken orally once per day over 12 weeks. Participants who achieved a clinical response after week 12 continued to take BMS-986165 12 mg orally once daily until the end of week 52. Participants who did not achieve clinical response prior to protocol v 3 but had an appropriate safety profile were eligible to receive BMS-986165 12 mg once per day. Participants who were randomized prior to the implementation of Protocol v3.0 who had not yet reached Week 12 but had an appropriate safety profile could switch to open-label BMS-986165 6 mg until week 52, if they did not achieve a clinical response at Week 12. Week 12 responders and week 12 non-responders who continued to derive a clinical benefit from their respective treatments at week 26/52 and week 52 respectively were eligible to receive open label BMS-986165 6 mg twice daily until week 104.
Period: Pre-Treatment Period
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Started | 60 | 86 | 84 | 9
Completed | 59 | 84 | 83 | 9
Not Completed | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other reasons | 1 | 1 | 1 | 0
Period: Treatment Period
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Started | 59 | 84 | 83 | 9
Completed | 13 | 14 | 14 | 4
Not Completed | 46 | 70 | 69 | 5
Not completed — Adverse Event | 11 | 20 | 18 | 2
Not completed — Lack of Efficacy | 18 | 12 | 13 | 2
Not completed — Withdrawal by Subject | 5 | 11 | 16 | 1
Not completed — Other reasons | 4 | 6 | 7 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 7 | 20 | 15 | 0
Not completed — Site terminated by sponsor | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165 | Total
Number analyzed (Participants) | 60 | 86 | 84 | 9 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (16.7) | 39.5 (15.2) | 37.9 (14.6) | 37.4 (13.7) | 38.8 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 38 | 34 | 3 | 97
  Male | 38 | 48 | 50 | 6 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 2 | 0 | 11
  Not Hispanic or Latino | 58 | 78 | 80 | 9 | 225
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Asian | 11 | 13 | 12 | 1 | 37
    Black or African American | 1 | 1 | 3 | 0 | 5
    White | 48 | 70 | 68 | 8 | 194
    Other | 0 | 2 | 0 | 0 | 2
    Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Achieving Clinical Remission at Week 12
Description: Percent of participants achieving clinical remission at Week 12. Clinical remission is defined as achieving a Crohn's Disease Activity Index (CDAI) Score below 150. CDAI is a tool that helps doctors measure how severe someone's Crohn's disease is. It uses questions about symptoms experienced over a week to calculate a score. The scores range from 0 to 600 and are classified into different categories. Scores from 0 to 149 suggest the disease may be in remission. Scores from 150 to 220 indicate mild activity. Scores from 220 to 450 mean the disease is moderate to severe. Scores from 451 to 600 indicate severe disease. Higher scores mean more severe symptoms.
  Risk Difference and Odds Ratio prespecified to be collected for 3 mg and 6 mg BMS-986165 arms only.
Time Frame: 12 weeks after first dose
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Number analyzed (Participants) | 60 | 86 | 84 | 9
Percent of Participants | 28.3 [16.9 to 39.7] | 32.6 [22.7 to 42.5] | 21.4 [12.7 to 30.2] | 22.2 [0.0 to 49.4]
Statistical Analysis 1: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — Cochran-Mantel-Haenszel stratified by geographic region (US, Japan, Rest of World), prior exposure to tumor necrosis factor inhibitor (TNFi; Exposed/Naive), and concomitant corticosteroid use (Yes/No); p = 0.5812, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = 4.3, 95% CI 2-sided [-11.0 to 19.5] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 2: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5812, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.6 to 2.5] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 3: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3720, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = -6.3, 95% CI 2-sided [-20.2 to 7.6] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 4: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3720, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 1.5] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)

2. Primary Outcome: Percent of Participants Achieving Endoscopic Response at Week 12
Description: Endoscopic Response is defined as >= 50% decrease from baseline in the Simple Endoscopic Score for Crohn's Disease (SES-CD). The SES-CD score is a way to measure how severe a person's bowel disease is. It looks at five different parts of the bowel and checks for things like ulcers and inflammation. Each part is given a score from 0 to 3 based on how bad the disease is. These scores are then added together for a total score ranging from 0 to 60. Higher scores indicate more severe disease. Baseline refers to the initial set of before data collected from participants before starting study treatment.
  Risk Difference and Odds Ratio prespecified to be collected for 3 mg and 6 mg BMS-986165 arms only.
Time Frame: 12 weeks after first dose
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Number analyzed (Participants) | 60 | 86 | 84 | 9
Percent of Participants | 8.3 [1.3 to 15.3] | 23.3 [14.3 to 32.2] | 16.7 [8.7 to 24.6] | 33.3 [2.5 to 64.1]
Statistical Analysis 1: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0198, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = 15.0, 95% CI 2-sided [3.7 to 26.3] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 2: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0198, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 3.4, 95% CI 2-sided [1.2 to 9.8] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 3: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1584, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = 8.2, 95% CI 2-sided [-2.6 to 19.0] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 4: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1584, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.7 to 6.1] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)

3. Secondary Outcome: Percent of Participants Achieving Clinical Response at Week 12
Description: Clinical response is defined as a reduction from baseline in the Crohn's Disease Activity Index (CDAI) score of ≥ 100 points or a total CDAI score < 150. CDAI is a tool that helps doctors measure how severe someone's Crohn's disease is. It uses questions about symptoms experienced over a week to calculate a score. The scores range from 0 to 600 and are classified into different categories. Scores from 0 to 149 suggest the disease may be in remission. Scores from 150 to 220 indicate mild activity. Scores from 220 to 450 mean the disease is moderate to severe. Scores from 451 to 600 indicate severe disease. Higher scores mean more severe symptoms. Baseline refers to the initial set of before data collected from participants before starting study treatment.
  Risk Difference and Odds Ratio prespecified to be collected for 3 mg and 6 mg BMS-986165 arms only.
Time Frame: 12 weeks after first dose
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Number analyzed (Participants) | 60 | 86 | 84 | 9
Percent of Participants | 40.0 [27.6 to 52.4] | 47.7 [37.1 to 58.2] | 38.1 [27.7 to 48.5] | 55.6 [23.1 to 88.0]
Statistical Analysis 1: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3464, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = 7.7, 95% CI 2-sided [-8.2 to 23.6] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 2: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3464, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.7 to 2.8] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 3: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8857, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = -1.2, 95% CI 2-sided [-17.0 to 14.7] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 4: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8857, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.5 to 1.9] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)

4. Secondary Outcome: Percent of Participants Who Achieving Patient Reported Outcomes 2 (PRO2) Remission at Week 12
Description: The Patient Reported Outcomes 2 (PRO2) is a way for patients to report how they're feeling. It focuses on two things: how often they have loose or liquid stools, and how much abdominal pain they have. They keep track of these things every day for a week. Stool frequency is rated on a scale from 0 to 3, with 0 being the normal number of stools per day to 3 which is >/=5 stools more than normal per day. The pain is rated on a scale from 0 to 3, with 0 being no pain and 3 being severe pain. The scores for these two things are added up to get a total score ranging from 0-6. If the average daily score for abdominal pain is 1 or less, and the average number of loose or liquid stools is 3 or less, then the disease might be in remission.
  Risk Difference and Odds Ratio prespecified to be collected for 3 mg and 6 mg BMS-986165 arms only.
Time Frame: 12 weeks after first dose
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Number analyzed (Participants) | 60 | 86 | 84 | 9
Percent of Participants | 25.0 [14.0 to 36.0] | 32.6 [22.7 to 42.5] | 20.2 [11.6 to 28.8] | 33.3 [2.5 to 64.1]
Statistical Analysis 1: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2841, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = 8.1, 95% CI 2-sided [-6.7 to 22.9] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 2: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2841, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.7 to 3.1] — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 3: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5417, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Risk Difference (RD) = -4.2, 95% CI 2-sided [-17.6 to 9.2] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 4: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5417, Mantel Haenszel — Based on a 2-sided test at a significance level of 0.025; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.3 to 1.8] — 6 mg BMS-986165 (numerator) vs Placebo (denominator)

5. Secondary Outcome: Change From Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12
Description: The SES-CD score is a way to measure how severe a person's bowel disease is. It looks at five different parts of the bowel and checks for ulcer size, ulcerated surface, inflamed surface, and stenosis. Each is given a score from 0 to 3 based on how bad the disease is. These scores are then added together for a total score ranging from 0 to 60. Higher scores indicate more severe disease. Baseline refers to the initial set of before data collected from participants starting study treatment.
Time Frame: 12 weeks after first dose
Population: All randomized participants with available baseline and week 12 SES-CD scores.
Measure: Mean (Standard Deviation); unit: Change in Score on a Scale
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165
Number analyzed (Participants) | 50 | 70 | 58 | 7
Change in Score on a Scale | -1.5 (4.3) | -2.5 (6.5) | -3.7 (5.5) | -5.6 (8.5)
Statistical Analysis 1: Comparison: 3 mg BMS-986165; Test type: Equivalence — Mean Change From Baseline; ANCOVA; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-4.3 to -1.8], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: Placebo vs 3 mg BMS-986165; Test type: Superiority — Adjusted means, 95% confidence intervals, and p-values are from an analysis of covariance model with factors for geographic region, prior exposure to tumor necrosis factor inhibitor, and concomitant corticosteroid use, and the baseline value as a covariate; p = 0.0428, ANCOVA — Based on a 2-sided test at a significance level of 0.025; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.7 to -0.1], Standard Error of Mean 0.92 — 3 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 3: Comparison: 6 mg BMS-986165; Test type: Equivalence — Mean Change from Baseline; ANCOVA; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-4.8 to -2.0], Standard Error of Mean 0.70
Statistical Analysis 4: Comparison: Placebo vs 6 mg BMS-986165; Test type: Superiority — [test comment as in outcome 5, analysis 2]; p = 0.0177, ANCOVA — Based on a 2-sided test at a significance level of 0.025; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-4.1 to -0.4], Standard Error of Mean 0.95 — 6 mg BMS-986165 (numerator) vs Placebo (denominator)
Statistical Analysis 5: Comparison: Placebo; Test type: Equivalence — Mean Change From Baseline; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.6 to 0.3], Standard Error of Mean 0.75
Statistical Analysis 6: Comparison: 12 mg BMS-986165; Test type: Equivalence — Mean Change from Baseline; ANCOVA; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-9.7 to -2.3], Standard Error of Mean 1.88

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization until study completion (assessed up to approximately 63 months). SAEs and Other AEs were assessed from first dose to 30 days after last dose of study therapy (assessed for an average of 11 months up to approximately 24 months).
Description: All-Cause Mortality represents all randomized participants. Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- 6 mg BMS-986165 - Open Label: Participants from the Placebo, 3 mg BMS-986165, and 6 mg BMS-986165 arms who did not achieve clinical response at week 12 but had an appropriate safety profile were eligible to receive open-label BMS-986164 6 mg twice per day until week 52. Week 12 responders and week 12 non-responders who continued to derive a clinical benefit from their respective treatments at week 26/52 and week 52 respectively were eligible to begin/continue to receive BMS986165 6 mg twice daily. Participants who were randomized to the 12 mg BMS-986165 arm prior to the implementation of Protocol v3.0 who had not yet reached Week 12 but had an appropriate safety profile could switch to open-label BMS-986165 6 mg if they did not achieve a clinical response at Week 12. Week 12 responders and week 12 non-responders from this arm who continued to derive a clinical benefit from their respective treatments at week 26/52 and week 52 respectively were eligible to receive open label BMS-986165 6 mg twice daily until week 104.
- 12 mg BMS-986165 - Open Label: Participants who took 12 mg BMS-986165 up to week 12/52 who did not achieve clinical response prior to protocol v 3 but had an appropriate safety profile were eligible to enter the open label period and received BMS-986164 12 mg once per day until week 104.
Arm/Group | Placebo | 3 mg BMS-986165 | 6 mg BMS-986165 | 12 mg BMS-986165 | 6 mg BMS-986165 - Open Label | 12 mg BMS-986165 - Open Label
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/86 | 0/84 | 0/9 | 0/161 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/59 | 11/84 | 5/83 | 2/9 | 15/161 | 1/6
Other Adverse Events (participants affected / at risk) | 33/59 | 55/84 | 55/83 | 7/9 | 86/161 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | 3 mg BMS-986165 (N=84) | 6 mg BMS-986165 (N=83) | 12 mg BMS-986165 (N=9) | 6 mg BMS-986165 - Open Label (N=161) | 12 mg BMS-986165 - Open Label (N=6)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 3 | 5 | 2 | 1 | 6 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Norovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Craniofacial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | 3 mg BMS-986165 (N=84) | 6 mg BMS-986165 (N=83) | 12 mg BMS-986165 (N=9) | 6 mg BMS-986165 - Open Label (N=161) | 12 mg BMS-986165 - Open Label (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 1 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 7 | 0 | 10 | 0
Aphthous ulcer (Gastrointestinal disorders) | 2 | 3 | 8 | 0 | 7 | 0
Crohn's disease (Gastrointestinal disorders) | 9 | 10 | 10 | 1 | 17 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 6 | 4 | 0 | 7 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 2 | 0 | 5 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2 | 0 | 2 | 0
Asthenia (General disorders) | 3 | 2 | 1 | 1 | 3 | 0
Pyrexia (General disorders) | 4 | 4 | 7 | 0 | 9 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 6 | 5 | 11 | 0 | 22 | 1
Folliculitis (Infections and infestations) | 0 | 5 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 5 | 0 | 12 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 9 | 5 | 3 | 11 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 6 | 1 | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 1 | 1 | 0
Headache (Nervous system disorders) | 4 | 6 | 5 | 0 | 4 | 0
Breast haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6 | 0 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 9 | 12 | 0 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 5 | 5 | 0 | 6 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Trial terminated because of lack of efficacy in the short term acute phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT03599622/Prot_SAP_000.pdf